CLINICAL TRIAL: NCT00677248
Title: A Phase II, Placebo-Controlled, Double-Blind, Randomised, 10-Week, Parallel-Group Study to Assess the Efficacy of Different Doses of KB2115 as Add on to Ezetimibe Treatment in Patients With Primary Hypercholesterolemia
Brief Title: LDL-Cholesterol Lowering Effect of KB2115 as Add on to Ezetimibe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karo Bio AB (Industry)
Responsible Party: Chief Medical Officer, Karo Bio AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-007831-24
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-05

CONDITIONS: Hypercholesterolemia
Keywords: Eprotirome; KB2115; dyslipidemia; hypercholesterolemia; hypertriglyceridemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Hypertriglyceridemia | interventions — Ezetimibe; 3-((3,5-dibromo-4-(4-hydroxy-3-(1-methylethyl)phenoxy)phenyl)amino)-3-oxopropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Ezetimibe and placebo
  Interventions: Drug: Ezetimibe and placebo
- 2 (Experimental): Eprotirome dose 1 and ezetimibe
  Interventions: Drug: Eprotirome and ezetimibe
- 3 (Experimental): Eprotirome dose 2 and ezetimibe
  Interventions: Drug: Eprotirome and ezetimibe
- 4 (Experimental): Eprotirome dose 3 and ezetimibe
  Interventions: Drug: Eprotirome and ezetimibe

INTERVENTIONS:
Drug: Ezetimibe and placebo — Placebo or three different doses of eprotirome added to ezetimibe treatment
  Arms: 1
Drug: Eprotirome and ezetimibe — Placebo or three different doses of eprotirome added to ezetimibe treatment
  Arms: 2; 3; 4

SUMMARY:
Eprotirome (KB2115) is a liver selective thyroid hormone that can induce hyperthyroidism in the liver, while an euthyroid state is preserved in the extrahepatic tissue. Eprotirome has in clinical trials demonstrated pronounced reduction of several independent risk factors for the development of atherosclerotic cardiovascular diseases.

The purpose of the study is to assess the efficacy and safety of KB2115 as add on therapy to ezetimibe following 10 weeks of exposure compared to placebo. The aim of the study is to assess efficacy (LDL-cholesterol lowering effects) and safety of KB2115 and to define a clinically relevant dose or dose range for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 75 years
* Patient with primary hypercholesterolemia with an LDL-cholesterol > 3.0 mmol/L
* At randomization, diet as instructed by the investigator during the last 4 weeks prior to randomization and willingness to follow these instructions throughout the study

Exclusion Criteria:

* History of somatic or psychiatric disease/condition, which may interfere with the objectives of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 10 weeks

SECONDARY OUTCOMES:
Triglycerides | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Kristensen, MD, PhD, Study Chair — Karo Bio AB
Locations (1):
- Karo Bio AB, Huddinge, Sweden